CLINICAL TRIAL: NCT01344226
Title: Clinical Outcomes and Evaluation of Lotemax (Loteprednol Ophthalmic Solution ) 0.5% QID for Treatment of Ocular Inflammation Associated With Cataract Surgery
Brief Title: Clinical Outcomes and Evaluation of Lotemax 0.5% in Treatment of Ocular Inflammation Associated With Cataract Surgery
Status: Completed | Type: Observational
Sponsor: Toyos Clinic (Other)
Responsible Party: Principal Investigator, Melissa Toyos, Principal Investigator, Toyos Clinic
Other Study IDs: MMC-2011A
Record Dates: First submitted 2011-04-27; First posted 2011-04-29 (Estimated); Results first posted 2018-10-22 (Actual); Last update posted 2018-10-22 (Actual); Status verified 2018-01

CONDITIONS: Pseudophakia; Inflammation
Keywords: steroid responder
MeSH Terms: conditions — Pseudophakia; Inflammation | interventions — Loteprednol Etabonate; Ophthalmic Solutions

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: loteprednol 0.5% ophthalmic solution — Lotemax to be used QID starting day of cataract surgery and 21 days after for total of 22 days.
  Other Names: Lotemax; loteprednol

SUMMARY:
Investigate the intraocular pressure(pressure inside the eye) of patients who are treated with Lotemax after undergoing cataract surgery.

DETAILED DESCRIPTION:
This is a single-center study to evaluate the clinical outcomes of Lotemax 0.5% for the treatment of Ocular inflammation associated with cataract surgery. Subjects will be screened from one to 21 days prior to initiation of dosing with the test article. Subjects who sign the informed consent document and meet all inclusion/exclusion criteria will be eligible to participate in this study. Subjects will instill one drop of Lotemax into the study (operative) eye QID for a maximum of 22 days. Dosing with test article will begin the day of surgery and for 21 days after surgery. Subjects will be seen for evaluation on Days 1, 7±1, and 21 ± 2 following surgery. Subjects will be seen for a follow-up visit on Day 42 ± 3 following surgery, about 21 days after their last dose of test article.

In addition to the test article regimen, subjects will receive Vigamox TID 3 days prior to surgery. Patients will receive one drop of Timoptic XE 0.5%, Zymaxid on the day of surgery. Postoperatively, patients will receive Vigamox TID for ten days and Bromday QD for 3 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female 18 years of age scheduled for unilateral cataract surgery (phacoemulsification or extracapsular) with posterior chamber intraocular lens implantation.
2. Agree not to have any other ocular surgery in the study or fellow eye for duration of study.
3. Have a BCVA of 20/200 or better in either eye.
4. Willing/able to return for all required study visits.
5. Willing/able to follow instructions from the study investigator and their staff.
6. Able to self-administer test article (or have a caregiver available to instill all doses of test article).
7. If woman capable of becoming pregnant, agree to have urine pregnancy test(must be negative) at agree to use a medically acceptable form of birth control during study and for at least one week prior to and after completion of the study.
8. Have read, understood, and signed the informed consent document approved by Sterling Institutional Review Board.
9. Have IOP ≥ 5mmHg and ≤ 22mmHg, (in study eye) with or without anti-glaucoma therapy at the pre-operative screening visit (if > 22mmHg, adjust following pachymetry).

Exclusion Criteria:

1. Have known hypersensitivity to Lotemax or to any component of the test article (including "procedural" medications such as anesthetic and/or fluorescein drops, dilating drops, etc.).
2. Have a known hypersensitivity to non-steroidal or steroidal anti-inflammatory drugs (NSAIDs).
3. Have intraocular inflammation (i.e. cells or flare in the anterior chamber as measured on slit lamp exam) in the study eye at the screening visit.
4. Have a known blood dyscrasia or bone marrow suppression, a diagnosis of uncontrolled/unstable peptic ulcer disease, inflammatory bowel disease, or ulcerative colitis, or any uncontrolled/unstable pulmonary, cardiac, vascular, autoimmune, hepatic, renal, or central nervous system disease.
5. Have used ocular, topical, or systemic steroids within 14 days or depot steroid 30 days prior to initiation of dosing with the test article or throughout the duration of the study. Note: use of an opioid during surgery (e.g., fentanyl) is allowed.
6. Have uncontrolled glaucoma or IOP >/= 27mmHg.
7. Have active corneal pathology noted in the study eye at the screening visit. Active corneal pathology is defined as corneal pathology that is non-stable, or greater than mild, or will compromise assessment of the safety or efficacy of treatment.
8. Are pregnant or nursing.
9. Have participated in any other study of an investigational drug or device within 30 days prior to randomization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male or Female 18 years of age scheduled for unilateral cataract surgery with intraocular implant.
Sampling Method: Non-Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2011-04; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Toyos, MD, Principal Investigator — Discover Vision Centers
Locations (1):
- Discover Vision Centers, Independence, Missouri, United States

REFERENCES:
- See also: Click on "Current Studies" — http://www.discovervision.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients in one location of one surgeon's clinic about to undergo cataract surgery were recruited from July 2011 to May 2013.
Pre-assignment Details: patients had to be off of steroids for 14 days with no depot steroid injection for 30 days
Groups:
- Patients Receiving Loteprednol 0.5% Qid Post Phacoemulsificati: Subjects instilled one drop of topical loteprednol 0.5% suspension qid into the operative eye four times daily for a maximum of 22 days. Dosing began on the day of surgery and continued for 21 days postoperatively.
Period: Overall Study
Arm/Group | Patients Receiving Loteprednol 0.5% Qid Post Phacoemulsificati
Started | 49
Completed | 41
Not Completed | 8
Not completed — Protocol Violation | 2
Not completed — Withdrawal by Subject | 3
Not completed — Lack of Efficacy | 3

BASELINE CHARACTERISTICS:
Groups:
- Patients Receiving Loteprednol 0.5% Qid Post Phacoemulsificati: patients received loteprednol 0.5% suspension for 21 days following surgery in addition to pre and postoperative standard of care
Arm/Group | Patients Receiving Loteprednol 0.5% Qid Post Phacoemulsificati
Number analyzed (Participants) | 49
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.93 (9.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 19
Region of Enrollment [Number; unit: participants]
  United States | 49

OUTCOME MEASURES:

1. Primary Outcome: Investigate Clinical Outcomes for Intraocular Pressure After Treatment With Lotemax (Loteprednol Ophthalmic Solution) 0.5% QID in Subjects Who Have Undergone Cataract Extraction With Posterior Chamber Intraocular Implantation.
Description: Evaluate intraocular pressure change in mm Hg from baseline in the first 6 weeks following cataract surgery in individuals treated with Lotemax (loteprednol ophthalmic solution) 0.5% QID after cataract extraction with posterior chamber intraocular implantation.
Time Frame: baseline to 6 weeks
Measure: Mean (Standard Error); unit: mm Hg
Arm/Group | Patients Receiving Loteprednol 0.5% Qid Post Phacoemulsificati
Number analyzed (Participants) | 49
mm Hg | -1.8 (1.06)

2. Secondary Outcome: ETDRS Letters Read Over Early Postoperative Period
Description: Final visual acuity at pod 42 as measured by ETDRS letters read was compared with baseline was measured for this outcome measure.
Time Frame: change in ETDRS letters read baseline to 6 weeks
Measure: Mean (Standard Error); unit: change in ETDRS letters read
Arm/Group | Patients Receiving Loteprednol 0.5% Qid Post Phacoemulsificati
Number analyzed (Participants) | 41
change in ETDRS letters read | 8.05 (2.14)

3. Secondary Outcome: Cell Scores in the Early Outcome Period as Measured at 6 Weeks Post Phacoemulsification
Description: Cell scores at the final visit (pod 42) will be compared with baseline cells and will be measured using 1mmx1mm slit lamp beam. White cells present in the anterior chamber in a 1mm x 1mm slit lamp beam measured 3 times with the average number of cells being recorded. The grading scale was 0 (no cells/high power field), 1 (1-5 cells/high power field), 2 (6-15 cells/high power field), 3 (16-25 cells/high power field) and 4 (>25 cells/high power field). Minimal values represent less inflammation or better inflammatory control and could represent a better outcome.
Time Frame: baseline to 6 weeks
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Patients Receiving Loteprednol 0.5% Qid Post Phacoemulsificati
Number analyzed (Participants) | 41
units on a scale | 0.25 (1.11)

4. Secondary Outcome: Flare Scores in Early Postoperative Period
Description: Flare scores will be measured using a 1mmx1mm slit lamp beam. Flare was assessed by looking at a 1mmx1mm slit lamp beam into the anterior chamber. Three measurements were taken and the average flare score was reported. The final outcome measure was the final flare score at 42 days compared to baseline. The grading scale was 0-4 with 0 repesenting no flare, 1mild flare, 2 moderate flare, 3 moderate severe and 4 severe flare. Minmal values represent less inflammation and could represent better inflammatory control.
Time Frame: baseline to 6 weeks
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Patients Receiving Loteprednol 0.5% Qid Post Phacoemulsificati
Number analyzed (Participants) | 41
units on a scale | 0.08 (0.78)

ADVERSE EVENTS:
Time Frame: 6 weeks after phacoemulsification was performed
Arm/Group | Patients Receiving Loteprednol 0.5% Qid Post Phacoemulsificati
Serious Adverse Events (participants affected / at risk) | 0/49
Other Adverse Events (participants affected / at risk) | 3/49
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patients Receiving Loteprednol 0.5% Qid Post Phacoemulsificati (N=49)
increasing ocular cell (Eye disorders) | 3 (3) — Patients exited from the study with increasing intraocular cells and/or pain requiring additional topical medications for inflammation. Subjective complaints and slit lamp exam were collected together at every scheduled and unscheduled visit.

LIMITATIONS AND CAVEATS:
Single surgeon, single site study with no randomization or masking. Fewer patients analyzed than anticipated due to competitive recruiting with similar studies.4 screen failures and 8 early terminations.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No